CLINICAL TRIAL: NCT02040714
Title: Multicenter Prospective Cohort Study on Current Treatments of Legg-Calvé-Perthes Disease
Acronym: IPSG1
Status: Enrolling by invitation | Type: Observational
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Collaborators: Alberta Children's Hospital (Other); Alfred I. duPont Hospital for Children (Other); Le Bonheur Children's Hospital (Other); Children's Hospital Colorado (Other); Children's Hospital Los Angeles (Other); Children's National Research Institute (Other); Children's Healthcare of Atlanta (Other); Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); Columbia University (Other); Connecticut Children's Medical Center (Other); Gillette Children's Specialty Healthcare (Other); Boston Children's Hospital (Other); Johns Hopkins University (Other); Kaiser Permanente (Other); Kasturba Medical College (Other); Montefiore Medical Center (Other); Nationwide Children's Hospital (Other); NYU Langone Health (Other); OrthoCarolina Research Institute, Inc. (Other); University of Sao Paulo General Hospital (Other); Seoul National University Childrens Hospital (Other); Shriners Hospitals for Children (Other); University Hospital Southampton NHS Foundation Trust (Other); Baylor College of Medicine (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); British Columbia Children's Hospital (Other); Children's of Alabama (Other); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); University of Oklahoma (Other); Oregon Health and Science University (Other); Rady Children's Hospital, San Diego (Other); San Jorge Children's Hospital (Puerto Rico) (Unknown); University College Dublin (Other); Tianjin Children's Hospital (Other); University Hospital Schleswig-Holstein (Other); University of California, San Francisco (Other); University of Haifa (Other); Uppsala University (Other); Medical University of Lodz (Other); Oslo University Hospital (Other); Seattle Children's Hospital (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Harry Kim, MD, Director of Research, Texas Scottish Rite Hospital for Children
Other Study IDs: IPSG 001
Record Dates: First submitted 2014-01-02; First posted 2014-01-20 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Legg Calve Perthes Disease
Keywords: femur head necrosis; hip; pediatric orthopedics; MRI; Osteonecrosis; Bone diseases; Legg Calve Perthes Syndrome
MeSH Terms: conditions — Legg-Calve-Perthes Disease; Femur Head Necrosis; Osteonecrosis; Bone Diseases | interventions — Osteotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (12):
- Nonoperative management between ages 6-8 in early stage: The choice of non-osteotomy management without containment or surgical containment would be solely governed by the current practice of the participating surgeons (i.e. the current practice of the individual surgeon would be followed within the broad framework of the study).
  Interventions: Procedure: Nonoperative Observation
- Operative management between age 6-8 in early stage: Operative containment treatment (femoral or pelvic osteotomy or Shelf acetabuloplasty) rendered in the early stage of the disease process
  Interventions: Procedure: Osteotomy + Long Term Non-Weight Bearing; Procedure: Osteotomy + Short Term Non-Weight Bearing
- Nonoperative management between age 8-11 in early stage: Patients who do not undergo some form of containment surgery because of medical, social, or other reasons will receive no surgical treatment.
  Interventions: Procedure: Nonoperative Observation
- Operative containment with short-term non-weightbearing in early stage: As per the current standard practice for patients between age 8-11 in developed countries, all patients will undergo some form of containment surgery (pelvic or femoral osteotomy) in order to better "contain" the femoral head underneath the acetabulum. Post-operative treatment will include 6 weeks of non-weight bearing on the operated leg.
  Interventions: Procedure: Osteotomy + Short Term Non-Weight Bearing
- Operative containment with prolonged non-weightbearing in early stage: As per the current standard practice for patients between age 8-11, all patients will undergo some form of containment surgery (pelvic or femoral osteotomy) in order to better "contain" the femoral head underneath the acetabulum. Post-operative treatment will include 6 months of non-weight bearing on the operated leg.
  Interventions: Procedure: Osteotomy + Long Term Non-Weight Bearing
- Operative containment for over 11 age group: Patients presenting over age 11 may receive multiple drilling and be non weight bearing for up to 6 months according to the treating physician's preference. Patients with application of fixator (arthrodiastasis) will be studied in this cohort arm as well, which typically involved 3-4 months followed by 8-12 weeks of non-weight bearing after fixator removal. Other surgical techniques may be included, however these are the most common for this age group.
  Interventions: Procedure: Osteotomy + Long Term Non-Weight Bearing; Procedure: Osteotomy + Short Term Non-Weight Bearing; Procedure: Multiple Epiphyseal Drilling
- Nonoperative management in over 11 age group: Patients will be non-weight bearing and receive physical therapy according to the physician preferences.
  Interventions: Procedure: Nonoperative Observation
- Nonoperative management in 1-6 age group: The choice of non-osteotomy management without containment or surgical containment would be solely governed by the current practice of the participating surgeons (i.e. the current practice of the individual surgeon would be followed within the broad framework of the study).
  Interventions: Procedure: Nonoperative Observation
- Operative management in 1-6 age group: The choice of osteotomy management with containment would be solely governed by the current practice of the participating surgeons (i.e. the current practice of the individual surgeon would be followed within the broad framework of the study).
  Interventions: Procedure: Osteotomy + Long Term Non-Weight Bearing; Procedure: Osteotomy + Short Term Non-Weight Bearing; Procedure: Multiple Epiphyseal Drilling
- Late Stage Bracing group: Patients presenting with <= 20 degrees of abduction on a maximum abduction x-ray treated with bracing who also present in the late stages of the disease (Waldenstrom Stage IIb or IIIa).The choice of management with or without containment or surgical containment would be solely governed by the current practice of the participating surgeons (i.e. the current practice of the individual surgeon would be followed within the broad framework of the study).
  Interventions: Procedure: Nonoperative Observation
- Late Stage Symptomatic treatment group: Patients presenting in the late stages of the disease (defined as Waldenstrom stage IIb or IIIa) who are treated symptomatically. The choice of management with or without containment or surgical containment would be solely governed by the current practice of the participating surgeons (i.e. the current practice of the individual surgeon would be followed within the broad framework of the study).
  Interventions: Procedure: Nonoperative Observation
- Late Stage Surgical Containment group: Patients presenting in the late stages of the disease (defined as Waldenstrom stage IIb or IIIa) who are treated with surgical containment. The choice of management with or without containment or surgical containment would be solely governed by the current practice of the participating surgeons (i.e. the current practice of the individual surgeon would be followed within the broad framework of the study).
  Interventions: Procedure: Osteotomy + Long Term Non-Weight Bearing; Procedure: Osteotomy + Short Term Non-Weight Bearing; Procedure: Multiple Epiphyseal Drilling

INTERVENTIONS:
Procedure: Osteotomy + Long Term Non-Weight Bearing — Surgical procedure that improves femoral head containment, plus a post-operative protocol that requires patient to maintain non-weight bearing for 6 months.
  Groups: Late Stage Surgical Containment group; Operative containment for over 11 age group; Operative containment with prolonged non-weightbearing in early stage; Operative management between age 6-8 in early stage; Operative management in 1-6 age group
Procedure: Osteotomy + Short Term Non-Weight Bearing — Surgical procedure that improves femoral head containment, plus a post-operative protocol that allows early return to function after 6 weeks of non-weight bearing.
  Groups: Late Stage Surgical Containment group; Operative containment for over 11 age group; Operative containment with short-term non-weightbearing in early stage; Operative management between age 6-8 in early stage; Operative management in 1-6 age group
Procedure: Nonoperative Observation — Group will not undergo any surgical or invasive procedures during course of treatment.
  Groups: Late Stage Bracing group; Late Stage Symptomatic treatment group; Nonoperative management between age 8-11 in early stage; Nonoperative management between ages 6-8 in early stage; Nonoperative management in 1-6 age group; Nonoperative management in over 11 age group
Procedure: Multiple Epiphyseal Drilling — Multiple epiphyseal drilling is a procedure that creates small holes in the femoral head growth plate to increase blood flow into the femoral head.
  Groups: Late Stage Surgical Containment group; Operative containment for over 11 age group; Operative management in 1-6 age group

SUMMARY:
Legg-Calvé-Perthes disease is a childhood hip disorder which is common enough to be a significant public health problem (affects 1 in 740 boys between ages 0-14), but uncommon enough to have a sufficient number of patients from a single institution to perform a definitive prospective study comparing the results of current treatments. The present study will establish a database of prospectively identified patients with Legg-Calvé-Perthes (LCP) Disease and collect information regarding their presentation, treatment, and outcomes in the course of receiving currently available treatments.

This study seeks to compare the outcomes of current treatments in the management of different age groups (ages 1-6, 6-8, 8-11, >11) of patients with Perthes disease at two- and five-year followup and at skeletal maturity. For each age group, two to three common treatment regimens currently used by practicing pediatric orthopaedic surgeons will be compared. The intervention a patient receives is determined through physician treatment expertise, and is not pre-determined by the study.

DETAILED DESCRIPTION:
Approximately 50 pediatric orthopaedic surgeons from pediatric centers in the US and other countries have agreed to participate in this database as members of the International Perthes Study Group (IPSG). TSRH will be the lead center. Sites who agree to participate will seek IRB approval from their own institutions. Data will be collected prospectively and entered into REDCap (Research Electronic Data Capture), a browser-based research database.

1-6 Cohort: For the 1-6 age patient group, patients involved in any treatment will be asked to participate in the study.

6-8 Cohort: For the 6-8 age patient group, patients presenting in an early stage of the disease (stage I or IIa), the surgeons who treat their patients with one of the following three treatment regimens currently used in practice will be asked to participate in the study :

1. Non-operative management (i.e., no osteotomy but can include soft tissue release);
2. Operative containment treatment (femoral or pelvic osteotomy or Shelf acetabuloplasty).

8-11 Cohort: For the 8-11 patient age group, patients presenting in an early stage of the disease (stage I or IIa), the surgeons who treat their patients with one of the following treatment regiments currently used in practice will be asked to participate in the study:

1. Non-operative management (i.e., no osteotomy);
2. Operative containment treatment (femoral or pelvic osteotomy or Shelf acetabuloplasty) followed by 6 weeks of postoperative non-weight bearing; and,
3. Operative containment treatment (femoral or pelvic osteotomy or Shelf acetabuloplasty) followed by 6 months of postoperative non-weight bearing.

>11 Cohort Registry: For the >11 patient age group, we will collect prospective data from surgeons who are currently treating their patients with any treatment regimens.

Patients who present to an IPSG member or their group during the late stages of the disease (stage IIb or stage III) will also be arranged into four separate age cohorts, identical to the list above. We will collect prospective data for these cases, as well.

Regardless of the patient's stage at enrollment, the patient's age at diagnosis or assigned cohort, the following data will be collected: information regarding patient characteristics at presentation, physical exam findings, responses to Perthes patient and/or outcomes questionnaires, and results of radiographic and MR imaging.

Participants will be assigned a unique study number. A secure web application, REDCap, will be used to capture and store research information including radiographic and MR images, clinical information, and de-identified outcomes questionnaire responses. Data will be transmitted and stored on a secure and dedicated server for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Legg-Calvé-Perthes disease
* Between age 1-18
* Patients with possible secondary femoral osteonecrosis if over the age of 11 due to trauma or corticosteroid therapy are also eligible.

Exclusion Criteria:

* Patients with previous surgical treatment on the affected hip

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with a recent diagnosis of Perthes disease that are being followed by a participating orthopedic surgeon. Participants are invited to participate during a visit to their treating hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-08; Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Sphericity deviation score of the femoral head | 5 years post intervention
  The primary outcome for each age group will be a quantitative estimate of the sphericity of the femoral head as a measure of femoral head deformity. A more deformed head will be less spherical. Greater deformity leads to an increased risk of arthritis early in life.

SECONDARY OUTCOMES:
Perfusion percentage | Just after diagnosis of Perthes disease
  The perfusion percentage is a measure of the amount of blood flow in the femoral head relative to the volume of the whole head. This measure is calculated from the perfusion MRI images that are collected just prior to the application of the intervention.

OTHER OUTCOMES:
Stulberg classification | at 2 years and 5 years post intervention
  The Stulberg classification is a categorical system used to describe the shape of the femoral head that is traditionally used to evaluate outcomes and arthritis risk for patients with Perthes disease.

CONTACTS AND LOCATIONS:
Overall Officials: Harry KW Kim, MD, MS, Study Chair — Texas Scottish Rite Hospital for Children
Locations (46):
- United States (28):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Kaiser Permanente Hospital, Los Angeles, California
  - Rady Children's Hospital California, San Diego, California
  - UCSF Benioff Children's Hospitals, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I. DuPont Hospital for Children of the Nemours Foundation, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Orthopaedics of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - NYU Langone/Hospital for Joint Disease, New York, New York
  - New York Presbyterian Hospital (Columbia Campus), New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - OrthoCarolina, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Tennessee-Campbell Clinic, Germantown, Tennessee
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Women and Children's Hospital of Adelaide, Adelaide, South Australia, Australia
- Universidade de São Paulo, São Paulo, Brazil
- Canada (2):
  - Alberta Children's Hospital, Division of Paediatric Surgery, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
- Tianjin Hospital Pediatric Orthopedics, Tianjin, China
- Germany (3):
  - Children's Hospital Hamburg-Altona, Hamburg
  - Hospital of Schleswig-Holstein, Lübeck
  - University Hospital of Schleswig-Holstein (Campus Lubeck), Lübeck
- Kasturba Medical College (KMC), Manipal, Udupi, Karnataka, India
- Children's Health Ireland at Temple Street, Dublin, Ireland
- Oslo University Hospital, Oslo, Norway
- Medical University of Lodz, Lodz, Poland
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Hospital Infantil Universitario Nino Jesus, Madrid, Spain
- Uppsala University, Uppsala, Sweden
- Centre hopsitalier universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (2):
  - Alder Hey Children's Hosopital (University of Oxford), Liverpool
  - Southampton Children's Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Patient enrolled in study will be deidentified (a specific ID will be assigned to participants) in each respective site, Each site will be in charge of entering their respective data in a main database. Data analysis of this collective data will be done mainly through the host site.

REFERENCES:
- See also: IPSG Website — http://www.perthesdisease.org